CLINICAL TRIAL: NCT06334965
Title: Multi-modal Characterisation of Hepatocellular Carcinoma (HCC) Treated With Targeted Radionuclide Therapy (TRT): Prospective Interventional Multicentre National Cohort
Acronym: OPERANDI-HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230279
Record Dates: First submitted 2024-02-05; First posted 2024-03-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Radioembolization
Keywords: transarterial radioembolization; 18F Choline PET-MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-MRI (Experimental): PET-MRI added in care pathway
  Interventions: Other: Simultaneous 18F-Choline PET-MRI

INTERVENTIONS:
Other: Simultaneous 18F-Choline PET-MRI — before first TARE administration (after work-up procedure) and one month after TARE administration

SUMMARY:
OPERANDI project aims to address unmet clinical needs in the current management of advanced-stage HCC treated with TARE by exploring new opportunities provided by imaging-based artificial intelligence (AI) and data augmentation, simultaneous PET-MRI imaging, and novel approaches to increase patient selection and TARE efficacy (genomic profiling, radiopotentiators, and new radionuclides). The research aim to identify predictive and early markers indicative of TARE effectiveness based on a large prospective cohort of HCC patients. This cohort will be used to uncover relevant predictive signatures within the morphological, functional, and molecular imaging data using novel imaging-based AI approaches with a new patient imaging pathway including simultaneous 18F-Choline PET-MRI.

Considering this global objective, the objective of this clinical research protocol is to provide clinical, molecular and imaging data in a prospective standardized study, notably by performing systematic pretherapeutic PET-MRI, in patients with HCC treated with TARE.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary malignant liver tumors, considered the sixth most common cancer and the third major cause of cancer-related death. Its worldwide incidence is expected to increase in the future. Additionally, it shows marked intertumor and intratumor heterogeneity at the microscopic and molecular levels, and there are currently no reliable imaging markers for predicting response to TARE.

TARE is a highly advanced treatment that consists in intra-arterial injection of radioactive microspheres. TARE is already approved for liver metastases and HCC in most countries. So, TARE for HCC, is part of the therapeutic Armamentarium exerting antitumor effects based on radio-biological (DNA damage) and immunological mechanisms. TARE using most currently 90Yttrium-labeled microspheres has proven its non-inferiority with better tolerance and better tumor response in comparison with systemic treatments in patients with HCC.

While highly promising, patient stratification and early identification of responders are currently insufficient due to the lack of pertinent imaging biomarkers, either non-invasive or invasive. Furthermore, prior therapy-induced DNA damages may lead to tumor resistance, therefore reducing TARE efficacy. Hence, the absence of a personalized treatment strategy is an unmet need for patients with HCC. This may result in survival disadvantage for non-responders, who could benefit otherwise from early treatment change, with expected more favorable outcomes.

Simultaneous PET-MRI: OPERANDI proposes a completely innovative and holistic approach via PET-MRI guided therapy. The research hypothesis is that simultaneous PET-MRI imaging provides more robust non-invasive predictive biomarkers than classical approach and better correlation between quantification internal of radiation therapy dosimetry and clinical outcomes than PET-CT. This requires technological development of PET-MRI, with most methodological challenges being attenuation correction, reducing the impact of organ motion due to respiration and cardiac motion, and minimizing truncation and susceptibility artifacts.

A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan. This new hybrid technology harnesses the strengths of PET and MRI to produce some of the most highly detailed images currently available. MRI scans use a strong (1.5 to 3T for clinical use) magnetic field to produce detailed morphologic images and some sequences provide functioning information (such as diffusion-weighted, dynamic contrast-enhanced, MR elastography sequence). PET scans use tracers according to the clinical indications to highlight metabolism changes. In HCC, the most common radiotracers are fluorodeoxyglucose (FDG) or Choline, which detect metabolically active malignant lesions.

OPERANDI project aims to address unmet clinical needs in the current management of HCC treated with TARE by exploring new opportunities provided by imaging-based artificial intelligence (AI) and data augmentation, simultaneous PET-MRI imaging, and novel approaches to increase patient selection and TARE efficacy (genomic profiling, radiopotentiators, and new radionuclides). Investigators aim to identify predictive and early markers indicative of TARE effectiveness based on a large prospective cohort of HCC patients. This cohort will be used to uncover relevant predictive signatures within the morphological, functional, and molecular imaging data using novel imaging-based AI approaches with a new patient imaging pathway including simultaneous PET-MRI.

Considering this global objective, the objective of this clinical research protocol is to provide clinical, molecular and imaging data in a prospective standardized study, notably by performing systematic pretherapeutic and follow-up PET-MRI, in patients with HCC treated with TARE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC for whom TARE decision was made at the MDT
* Patients ≥ 18 years of age
* Diagnosis of HCC based on imaging (EASL guidelines) and confirmed histologically
* At least one target lesion to be treated by radioembolisation, naïve to any previous treatment
* Child-Pugh Class < B8
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy ≥ 3 months
* Available baseline imaging (multiphasic CT), performed within 6 weeks before the beginning of TARE

Exclusion Criteria:

* Patient with contraindication to MRI
* Patient with contraindication to 18F-choline : potential hypersensitivity to the product or to any excipients
* Non-adequate bone marrow, liver and renal function within 15 days prior to work-up as assessed by the following laboratory tests:

  * Hemoglobin ≤ 8.0 g/Dl
  * Platelet count < 50,000/ mm3
  * Total bilirubin > 3 mg/dL (or > 51 µmol/ L).
  * Prothrombin time ≤ 50%
  * Glomerular Filtration Rate (GFR) < 35 mL/min/1.73 m2
* Infiltrating tumor more than 70% of the liver
* Prior liver transplantation
* Initial prescription for SIRT and concomitant systemic treatment
* Patient refusal to give written and informed consent
* No affiliation to a social security regimen or CMU
* Patient under State Medical Aid
* Known pregnancy or breastfeeding women
* Patient deprived of freedom, subject under a legal protective measure
* Any significant medical, psychiatric, or surgical condition that is uncontrolled and could endanger the subject's safety or limit adherence to the study's objectives and assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Clinical response | 12 months after the day of first administration of TARE
  Clinical response defined by the PFS as the time measured from the day of first administration of TARE to first progression or death at 12 months, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Catherine ANSQUER, Dr, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - Service de Médecine Nucléaire, Hôpital Beaujon, Clichy
  - Beaujon hospital, Clichy
  - CHU Nantes, Nantes
  - Service de Médecine Nucléaire, CHU de Nantes, Nantes
  - Service de medecine nucleaire, Hôpital Bichat, Paris

IPD SHARING:
Plan to Share IPD: No